CLINICAL TRIAL: NCT04915937
Title: Tolerance of Term Infants Fed Formula With Oligosaccharides
Brief Title: Formula Tolerance of Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AL41
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Gastro-Intestinal Tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Infant Formula (Experimental): Feed ad libitum during study period
  Interventions: Other: Study Infant Formula

INTERVENTIONS:
Other: Study Infant Formula — RTF milk-based infant formula with oligosaccharides

SUMMARY:
To assess the effects of infant formula with oligosaccharides on symptoms of formula intolerance in healthy, term infants

ELIGIBILITY:
Inclusion Criteria:

* Participant is judged to be in good health as determined from participant's medical history by parent report
* Participant is a singleton from a full-term birth with a gestational age of 37-42 weeks.
* Participant's birth weight was >= 2490 g (~5 lbs. 8 oz.)
* Participant was identified by parents as very fussy or extremely fussy in the Baseline Tolerance Evaluation on a formula-feed
* Participant is exclusively formula-fed at time of study entry and Parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study, unless instructed otherwise by their healthcare professional.
* Parent(s) confirm their intention not to administer vitamin, mineral, human milk oligosaccharide(s) (HMO), prebiotic(s), or probiotic(s) supplements (with the exception of vitamin D supplements if instructed by their healthcare professional), non-study formula, foods, juices, or other sources of nutrition to their infant from enrollment through the duration of the study
* Participant's parent(s) has voluntarily signed and dated an Informed Consent Form (ICF), approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC) and provided applicable local privacy regulation authorization prior to any participation in the study

Exclusion Criteria:

* An adverse maternal, fetal, or participant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development. This includes but is not limited to suspected maternal substance abuse.
* Participant is taking and plans to continue taking medications (including OTC, such as Mylicon® for gas), home remedies (such as juice for constipation), herbal preparations, or rehydration fluids that might affect GI tolerance.
* Participant participates in another study that has not been approved as a concomitant study
* Participant has been fed a formula with greater than 2 HMOs prior to study enrollment
* Participant has been fed an extensively hydrolyzed, amino acid based, or preterm formula within 14 days prior to study enrollment and/or an extensively hydrolyzed, amino acid based, or preterm formula has been recommended by the physician.
* Participant has an allergy or intolerance to any ingredient in the study product, as reported by the parent
* Participant has been treated with antibiotics within 7 days prior to enrollment

Ages: 7 Days to 65 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Fussiness | Baseline to Study Day (SDAY) 2
  Absolute and % change in fussiness severity reported from Daily Tolerance Diary

SECONDARY OUTCOMES:
Gastrointestinal Tolerance | Baseline to SDAY 28
  Parent Completed Diary
Stool | Baseline to SDAY 28
  Parent Completed Diary

OTHER OUTCOMES:
Formula Intake | SDAY 1 to SDAY 28
  Parent Completed Diary
Weight | SDAY 1 to SDAY 28
  Weight gains, percentiles, and z-scores
Length | SDAY 1 to SDAY 28
  Length gains, percentiles, and z-scores
Infant Feeding and Stool Patterns Questionnaire | SDAY 1 and SDAY 28
  Parent completed questionnaire; 16, 5-point Likert scale questions, scaled from frequent to less frequent
Formula Satisfaction Questionnaire | SDAY 1 and SDAY 28
  Parent completed questionnaire; 13 questions of up to 5 categories scaled from positive to negative
Parental perspectives | SDAY 1 and SDAY 28
  Parent completed questionnaire; 4, 5-point Likert scale questions, scaled from negative to positive
Health Resource Utilization | SDAY 7 and SDAY 28
  Number of Visits
Adverse Events | SDAY 1 to SDAY 28
  Standard adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Reverri, PhD, MS, RD, Study Chair — Abbott Nutrition
Locations (12):
- United States (12):
  - MedPharmics, LLC, Phoenix, Arizona
  - Dade Research Center, LLC, Miami, Florida
  - Meridian Clincial Research- Macan, Macon, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Springs Medical Research, Owensboro, Kentucky
  - MedPharmics, Covington, Louisiana
  - Boeson Research Kalispell, Kalispell, Montana
  - Meridian Clinical Research, Hastings, Nebraska
  - Be Well Clinical Studies, Lincoln, Nebraska
  - AVIATI Healthcare & Clinical Research, Memphis, Tennessee
  - Invesclinic US LLC, Edinburg, Texas
  - Maximos Ob/Gyn, League City, Texas

IPD SHARING:
Plan to Share IPD: No